CLINICAL TRIAL: NCT06632496
Title: BD Prevue(TM) II Peripheral Vascular Access System With Cue(TM) Needle Tracking Technology Clinical Study
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-23PREVUE001
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: BD Prevue II for Peripheral Intravenous Catheter Placement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- USGPIV: Patient who is a candidate for an ultrasound-guided peripheral intravenous catheter (USGPIV) placement procedure (midline catheters included) using BD Prevue(TM) II Peripheral Vascular Access System with Cue(TM) Needle Tracking Technology as assessed per their clinician(s)
  Interventions: Device: BD Prevue(TM) II

INTERVENTIONS:
Device: BD Prevue(TM) II — Ultrasound-guided peripheral intravenous catheter placement procedure using the BD Prevue(TM) II

SUMMARY:
This post-market study is being conducted to generate safety and performance data on the BD Prevue(TM) II Peripheral Vascular Access System with Cue(TM) Needle Tracking Technology. The data will be utilized to support regional registrations (for example, EU MDR), and document any unforeseen residual risks.

DETAILED DESCRIPTION:
This is an observational post-market, human subject study to evaluate the safety and performance of the BD Prevue(TM) II Peripheral Vascular Access System with Cue(TM) Needle Tracking Technology. Subjects will be recruited for participation based on need for IV catheter (midline catheters included) placement in a hospital setting.

Enrolled subjects will go through ultrasound-guided peripheral intravenous catheter (USGPIV) placement as part of their clinical care. USGPIV is defined as a procedure in which an ultrasound machine is used to assist a qualified health care provider with IV cannulation from skin puncture through venipuncture via direct visualization on the ultrasound machine in real time.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 years, or older
* A patient who is a candidate for an ultrasound-guided peripheral intravenous catheter (midline catheters included) placement procedure using BD PrevueTM II Peripheral Vascular Access System with CueTM Needle Tracking Technology as assessed per their clinician(s)
* Able and willing to provide informed consent or legal authorized representative (LAR) authorized to give consent on behalf of the subject

Exclusion Criteria:

* Any patient in whom ultrasound procedure might interfere with medical care or create undue hardship
* Known, or suspected, allergy to materials contained in the BD PrevueTM II Peripheral Vascular Access System with CueTM Needle Tracking Technology or accessories that may come in contact with the patient
* Localized skin, tissue, or other clinical factors that would prevent completion of the ultrasound procedure
* Previous medical history that would prevent completion of the ultrasound procedure

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are defined as patients who need to receive insertion of a peripheral IV (midline catheters included) catheter as part of their medical treatment
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Primary Performance: To provide visualization of the target vessel in which to insert the chosen vascular access device | During the procedure
  The PrevueTM II system is able to visualize the target vasculature (>=70% with a 95% confidence interval)
Primary Performance: To have successful vascular access either by cannulation or blood return. | During the procedure
  Successful access with the vascular access device, either by cannulation or blood return (>=70% with a 95% confidence interval)
Primary Performance: To determine if BD Prevue(TM) II Peripheral Vascular Access System with Cue(TM) Needle Tracking Technology is able to provide visual needle tip location tracking to assist with insertion of the chosen vascular access device. | During the procedure
  CueTM Needle Tracking System is able to properly display the location of the needle tip during vascular access device access insertion (>=80% with a 95% confidence interval)
Primary Safety: To determine the incidence of device related adverse events, experienced by patient or user, when using the BD PrevueTM II Peripheral Vascular Access System with CueTM Needle Tracking Technology | During the procedure and 15 minutes after the procedure
  Rate of device related adverse events (<2%).

SECONDARY OUTCOMES:
Secondary Performance: To have successful first-attempt vascular access either by cannulation or blood return when using the BD PowerGlide Pro midline catheter. | During the procedure
  Successful first-attempt access with the PowerGlide Pro midline catheter, either by cannulation or blood return (>=70% with a 95% confidence interval)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brookdale University Hospital & Medical Center, Brooklyn, New York
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No